CLINICAL TRIAL: NCT04851678
Title: Longitudinal Impact of Stressors in Adults With Tourette Syndrome
Acronym: LISA-TS
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David Isaacs, Assistant Professor, Neuro-Movement Disorders Division, Vanderbilt University Medical Center
Other Study IDs: U12134
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Tourette Syndrome
Keywords: Stress; Environmental stress; Psychosocial stress
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with Tourette syndrome (TS): Individuals previously diagnosed with Tourette syndrome (TS). Participants must be 18 years of age or older.
  Interventions: Other: None - observational study

INTERVENTIONS:
Other: None - observational study — None - observational study

SUMMARY:
The Investigators propose a two-year, longitudinal pilot study of TS adults (>18) to determine impact of lifetime environmental stress exposure on tic severity, psychiatric comorbidity severity, and health-related quality of life (HRQOL).

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a widely prevalent neurodevelopmental disorder with limited treatment options,(1,2) substantial impact on quality of life in children(3-7) and adults,(4,8-10) and two-fold increased risk of premature death.(11,12) Tics are the defining feature of TS, and as a result, TS is often narrowly perceived in terms of tics alone. Tics themselves tend to wane in late adolescence, with distressing tics persisting in only one-third of TS patients.(13) Because tics generally diminish with age, the plight of adults with TS is often neglected. Over half of TS adults suffer from anxiety and depression,(10,14) and a similar percentage experience symptoms of attention deficit hyperactivity disorder (ADHD) and obsessive-compulsive disorder (OCD), findings recently corroborated in our own clinical population.(10) Many TS adults struggle to form meaningful relationships with peers, and one-third feel inadequately supported by their families.(13) The burden of TS in adulthood extends beyond mental and social health. In a national registry cohort study, individuals with TS had a mortality rate ratio of 1.8 relative to healthy controls, even after controlling for comorbid psychiatric diagnoses.(11) The causes of more frequent premature death in TS populations are unclear, with many mechanisms implicated, including suicide,(15) traumatic accidents,(12) substance abuse,(16) metabolic disorders,(12,17) and complications from pharmacotherapy.(18,19)

Environmental stressors are also postulated to impact the course of TS.(20) An environmental stressor is any external condition or event that poses a threat to an individual's well-being.(21) Such stressors are known to alter brain development(22-24) and increase risk of adulthood psychopathology.(25,26) A single study has explored the role of environmental stressors in TS, finding that selected stressors predicted two-year tic and psychiatric symptom severity in a pediatric cohort (n=37 patients).(27) No similar investigations have been undertaken in TS adults. The Investigators hypothesize that environmental stressors are risk factors for more severe adult TS phenotype. The Investigators propose a two-year, longitudinal pilot study of TS adults (>18) to determine impact of lifetime environmental stress exposure on tic severity, psychiatric comorbidity severity, and health-related quality of life (HRQOL).

Aim 1. Determine influence of lifetime environmental stressors on tic severity in TS adults. Hypothesis: Number of lifetime stressors at baseline assessment is associated with greater tic severity at two year follow-up. Seventy adults with TS will be recruited from the Vanderbilt TS Clinic to complete a baseline assessment, consisting of validated clinical rating scales for tic severity (Yale Global Tic Severity Scale), common psychiatric comorbidities, and lifetime environmental stressors (Stress and Adversity Inventory for Adults, STRAIN). Because acute and chronic stressors exert differential physiologic and clinical-level effects,(28-31) the STRAIN assesses these separately. The Investigators will use multivariable linear regression to examine the influence of acute and chronic lifetime stressor count at baseline on tic severity at two years, controlling for baseline tic severity and psychiatric comorbidities, as well as anti-tic medications at follow-up. Results will clarify the impact of environmental stressors on tic severity in TS adults.

Aim 2. Determine influence of lifetime environmental stressors on depression in TS adults.

Hypothesis: Number of lifetime stressors at baseline assessment is associated with more depressive symptoms at two-year follow-up. Depression is the psychiatric symptom that most impacts adult functioning and QOL.(10) As part of baseline and follow-up assessments, Aim 1 participants will complete standardized, semi-structured psychiatric interviews (Mini International Neuropsychiatric Interview, MINI) and validated self-report depression scales (NeuroQOL-Depression). The statistical approach from Aim 1 will be adopted to examine the influence of acute and chronic lifetime stressor count at baseline on depression symptom severity at two years, again controlling for select confounds. Findings will delineate the effects of acute and chronic environmental stressors on depression in adults with TS.

Aim 3. Determine influence of positive childhood experiences on health-related quality of life (HRQOL) in TS adults. Hypothesis: Greater number of positive childhood experiences is associated with better HRQOL in TS adults at two-year follow-up. Positive childhood experiences partially mitigate the negative effects of adverse childhood experiences.(32) At baseline and follow-up visits, Aim 1 participants will report number and type of positive childhood experiences. They will also complete a validated HRQOL measure specific to TS: the Gilles de la Tourette-Quality of Life Scale (GTS-QOL). The Investigators will use multivariable regression modeling to examine the influence of positive childhood experiences on future HRQOL, controlling for environmental stressors and baseline HRQOL. Results will elucidate the potentially moderating role of positive childhood experiences on HRQOL in TS adults.

ELIGIBILITY:
Inclusion Criteria:

* adults (>18) meeting Diagnostic and Statistics Manual, 5th edition (DSM-V) criteria for Tourette syndrome, chronic motor tic disorder, or chronic vocal tic disorder
* ability to provide informed consent
* English proficiency

Exclusion Criteria:

- significant medical, neurologic, or psychiatric diagnoses (e.g. uncontrolled epilepsy, chronic heart failure, schizophrenia) besides TS and its commonly co-occurring psychiatric diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults (>18 years of age) with Tourette syndrome or other chronic tic disorder
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Tic Score from Yale Global Tic Severity Scale (YGTSS) | 2 years post-baseline assessment
  Semi-structured, clinician-administered interview to assess tic severity. Total tic scores are a composite of motor tic scores (0-25) and phonic tic scores (0-25) based on 5 dimensions of tic severity: number, frequency, intensity, complexity, and interference. Total tic scores range from 0-50. Higher scores indicate great tic severity. The YGTSS is the gold-standard clinical rating scale for tic severity.
NeuroQOL-Depression Score | 2 years post-baseline assessment
  NeuroQOL-Depression is a validated, 8-item self-report scale assessing symptoms of depression. Raw total scores range from 8-40; raw scores are converted to T-scores based on normative samples. Higher scores indicate more depressive symptoms. NeuroQOL-Depression is part of the Neuro-QOL (Quality of Life in Neurological Disorders) measurement system. The scale is designed to be completed with one minute.
Gilles de la Tourette Quality of Life Scale (GTS-QOL) Score | 2 years post-baseline assessment
  The GTS-QOL is a 27-item self-report scale. Respondents rate each item on a Likert scale ranging from 0 ("no problem") to 4 ("extreme problem"). The scale is composed of four sub-scales: Psychological (11 items), Physical/Activities of Daily Living (Physical/ADL) (7 items), Obsessive-Compulsive (OC) (5 items), and Cognitive (4 items) (39). Item scores within each subscale are summed and then normalized to 100 to generate the subscale score. The four subscale scores are then summed and normalized to 100 to yield the total score. Higher scores indicate worse health-related quality of life.

SECONDARY OUTCOMES:
NeuroQOL-Anxiety Score | 2 years post-baseline assessment
  NeuroQOL-Depression is a validated, 8-item self-report scale assessing symptoms of anxiety. Raw total scores range from 8-40; raw scores are converted to T-scores based on normative samples. Higher scores indicate more anxiety symptoms. NeuroQOL-Anxiety is part of the Neuro-QOL (Quality of Life in Neurological Disorders) measurement system. The scale is designed to be completed with one minute.
Adult ADHD Self-Report Screening Scale for DSM-V (ASRS-V) Score | 2 years post-baseline assessment
  ASRS-V is a 6-question scale screening for symptoms of inattention and hyperactivity. Each item is rated 0 ("never") to 4 ("very often"). Total score is the sum of individual item scores. Higher score indicates more ADHD symptoms. In clinical populations, ASRS-V total score cutoff ≥ 14 is 81% sensitive and 70% specific for detecting ADHD.
Dimensional Obsessive-Compulsive Scale (DOCS) Score | 2 years post-baseline assessment
  DOCS is a 20-item, validated self-report scale assessing for severity of obsessive-compulsive symptoms. Total score ranges from 0-80, with higher scores indicating more OCD symptoms. In clinical populations, DOCS total score cutoff ≥ 21 is 70% sensitive and 70% specific in distinguishing OCD from other anxiety disorders.

CONTACTS AND LOCATIONS:
Overall Officials: David A Isaacs, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided